CLINICAL TRIAL: NCT01095341
Title: Postoperative Hyperthyroidism After Parathyroidectomy
Brief Title: Postoperative Hyperthyroidism
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Priv. Doz. Dr. med. habil. Gottfried Rudofsky, University Hospital Heidelberg
Other Study IDs: GR-2010
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Hyperthyroidism
Keywords: hyperthyroidism; tertiary hyperparathyroidism; palpation thyroiditis; parathyroidectomy; thyroglobulin; rate of postoperative hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- THP: THP: patients undergoing parathyroidectomy according to tertiary hyperparathyroidism
  Interventions: Other: No intervention performed
- Other causes: patients with hyperthyroidism not caused by parathyroidectomy
  Interventions: Other: No intervention performed

INTERVENTIONS:
Other: No intervention performed

SUMMARY:
The purpose of this study is to evaluate the frequency and the clinical course of postoperative hyperthyroidism following surgery of tertiary hyperparathyroidism (THP) and to determine the diagnostic value of thyroglobulin in this setting.

ELIGIBILITY:
Inclusion Criteria:

* patients with tertiary hyperparathyroidism undergoing surgery for this reason
* dialysis treatment

Exclusion Criteria:

* patients wish

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with tertiary hyperparathyroidism undergoing surgery for this reason
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Hyperthyroidism

SECONDARY OUTCOMES:
Thyroglobulin elevation

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried Rudofsky, MD, Principal Investigator — University Hospital Heidelberg Germany
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Rudofsky G Jr, Grafe IA, Metzner C, Leowardi C, Fohr B. Transient post-operative thyrotoxicosis after parathyroidectomy. Med Sci Monit. 2009 Mar;15(3):CS41-3. PMID 19247247